CLINICAL TRIAL: NCT04123847
Title: Task-specific Epidural Stimulation and Training for Recovery of Stepping, Standing and Voluntary Movement Following Severe Spinal Cord Injury
Brief Title: Standing, Stepping and Voluntary Movement Spinal Cord Epidural Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Harkema PhD (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor-Investigator, Susan Harkema PhD, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17.1024 MC-PP-2
Record Dates: First submitted 2019-05-30; First posted 2019-10-11 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
Keywords: epidural stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Stand, Step and Voluntary Training (Experimental)
  Interventions: Other: Standing and Stepping; Device: Standing, Stepping and Voluntary Movement with spinal cord Epidural Stimulation

INTERVENTIONS:
Other: Standing and Stepping — Participants will have at least 80 sessions of stand and step training with the assistance of trainers over-ground, or in a harness on a body weight supported treadmill.
Device: Standing, Stepping and Voluntary Movement with spinal cord Epidural Stimulation — Participants will be have at least 80 sessions of stand and step training with epidural stimulation, with the assistance of trainers over-ground, or in a harness on a body weight supported treadmill. Voluntary movement with epidural stimulation will be completed in the supine or seated position.
  Other Names: Stand-scES; Step-scES; Vol-scES

SUMMARY:
This study will determine the level of functional gain, below the injury for voluntary control of movements, and recovery standing and stepping function as a result of activation of spinal circuits with scES in humans with severe paralysis. Training will consist of practicing stepping, standing and voluntary movements in the presence of specific scES configurations designed specific for stepping (Step-scES), specific for standing (Stand-scES) and for the voluntary movements of the legs and trunk (Vol-scES). Ability to step, stand, move voluntarily, as well as cardiovascular, respiratory, bladder, bowel and sexual function will be assessed in these individuals with chronic severe spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* non-progressive SCI
* at least 2 years post injury
* stable medical condition
* inability to walk independently overground
* unable to voluntarily move all individual joints of the legs

Exclusion Criteria:

* ventilator dependent
* untreated painful musculoskeletal dysfunction, fracture or pressure sore
* untreated psychiatric disorder or ongoing drug abuse
* cardiovascular, respiratory, bladder, or renal disease unrelated to SCI
* pregnant at the time of enrollment or planning to become pregnant during the time course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2025-11-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of lower extremity independence time during 10 min standing bout after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  We will measure the amount of time individuals are able to stand without manual assistance (independently) throughout a 10 min bout
Change from baseline of stepping independence time during 6 min stepping bout after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  We will measure the number of steps individuals are able to take without manual assistance (independently) throughout a 6 min stepping bout
Change from baseline of number of consecutive hip flexion repetitions performed within one minute after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  We will measure the ability of the individuals to perform consecutive hip flexion repetitions with stimulation during a 1-minute period

SECONDARY OUTCOMES:
Change from baseline in resting metabolic rate after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Resting metabolic rate
Change from baseline in forced vital capacity (FVC) after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Respiratory Motor Control Assessment
Change from baseline in maximum inspiratory pressure (MIP) after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Respiratory Motor Control Assessment
Change from baseline in forced expiratory volume in one second (FEV1) after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Respiratory Motor Control Assessment
Change in baseline in maximum expiratory pressure (MEP) after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Respiratory Motor Control Assessment (RMCA)
Change from baseline in bladder capacity after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using urodynamics we will measure bladder capacity in mL.
Change from baseline in bladder voiding efficiency after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using urodynamics we will measure voiding efficiency (leak amount/total capacity)x100.
Change from baseline in detrusor pressures during filling after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using urodynamics we will measure detrusor pressure in cmH2O.
Change from baseline in bladder compliance after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using urodynamics we will measure bladder compliance in mL/cmH2O.
Change from baseline in mean resting anal pressure after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using anorectal manometry we will measure mean resting pressure in mmHg.
Change from baseline in mean squeeze pressure after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using anorectal manometry we will measure mean squeeze pressure in mmHg.
Change from baseline in mean squeeze increase pressure after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using anorectal manometry we will measure mean squeeze increase pressure in mmHg.
Change from baseline in squeeze anal canal length after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using anorectal manometry will measure squeeze anal canal length in cm.
Change from baseline in bowel sensation after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  Using anorectal manometry we will measure bowel sensation in mL.
Change in baseline in sexual function after 160 sessions (1 year) | Baseline, 160 sessions (1 year)
  We will measure change in sexual health function using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Harkema, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No